CLINICAL TRIAL: NCT03507088
Title: Fluorine-18 Fluoroestradiol Positron Emission Tomography-computed Tomography: an in Vivo Biomarker Predicting Response to Fulvestrant in Women With Estrogen Positive Metastatic Breast Cancer?
Brief Title: Study to Determine the Utility of FES-PET in the Prediction of Response to Fulvestrant in Women With Estrogen Positive Metastatic Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhimin Shao (Other)
Responsible Party: Sponsor-Investigator, Zhimin Shao, professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1503144-6
Record Dates: First submitted 2018-04-03; First posted 2018-04-24 (Actual); Last update posted 2019-05-08 (Actual); Status verified 2019-05

CONDITIONS: Metastatic Breast Cancer
Keywords: fulvestrant 500 mg; fluorine-18 fluoroestradiol PET-CT
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All patients will undergo FES-PET/CT at baseline and FES-PET after 28 days of fulvestrant treatment. Whenever possible, tumor biopsies will be performed to correlate to FES-PET results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- fulvestrant (Experimental): 500mg fulvestrant on days 0, 14, 28 and every 28 days thereafter Fluoroestradiol-PET is performed at baseline and after 28 days
  Interventions: Drug: Fluoroestradiol (18F)

INTERVENTIONS:
Drug: Fluoroestradiol (18F) — A FES-PET/(CT) will be performed twice during protocol execution. Patients will be injected with approximately 222 MBq 18F-FES each time.

SUMMARY:
Effects of fulvestrant on the ERs may be evaluable by molecular imaging using positron emission tomography with the ER-specific FES tracer. In this study we will determine the utility of FES-PET in the prediction of response to fulvestrant 500 mg in women with estrogen positive metastatic breast cancer

DETAILED DESCRIPTION:
More than 70% of patients with metastatic breast cancer present with hormone receptor positive disease and for whom hormonal therapy is the preferred treatment approach. First-line treatment recommendations for women with hormone receptor positive locally advanced or metastatic disease includes a generation aromatase inhibitors or tamoxifen. Fulvestrant, a 17β-estradiol analog, is an antiestrogen that suppresses estrogen signaling by binding to ER and inducing oestrogen receptor degradation and has estrogen antagonistic activity but no estrogen agonistic effect. Fulvestrant has been shown to have superiority over other endocrine therapy in a series of randomized controlled trials.

The whole-body imaging of the availability of ER using FES-PET may prove valuable to evaluate the effects of fulvestrant on the ER non-invasively in individual patients. This potentially allows early prediction of therapy efficacy to fulvestrant in women with estrogen positive metastatic breast cancer.

In this pilot-study we will evaluate 35 patients who received fulvestrant as treatment for metastatic breast cancer. All patients will undergo FES-PET/CT at baseline and FES-PET after 28 days. Whenever possible, tumor biopsies will be performed to correlate to FES-PET results.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a history of histological proven ER-positive primary breast cancer and, whenever available, histological proven ER-positive recurrence.
2. No previous fulvestrant treatment
3. ER-antagonists should be discontinued for 5 weeks prior to FES-PET. The use of aromatase inhibitors is allowed.
4. Age > 18
5. ECOG 0-2
6. Life expectancy > 6 months
7. Informed consent obtained
8. Able to comply with the protocol

Exclusion Criteria:

1. Presence of life-threatening visceral metastases
2. Evidence of central nervous system metastases
3. > 3 lines of endocrine therapy for metastatic disease
4. Isolated liver metastasis (high FES uptake by normal liver)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
To evaluate the accuracy of the change of FES uptake in predicting progression-free survival(PFS) in patients treated with fulvestrant 500 mg | baseline; 28 days
  The FES-uptake will be calculated for all tumor lesions in individual patient at baseline and 28 days. Therapy response will be monitored by regular follow-up. RECIST criteria and clinical benefit will be used as criteria. All patients will be followed up until disease progression.

SECONDARY OUTCOMES:
Evaluate the heterogeneity of ER among different metastatic sites in breast cancer patients in vivo | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zhiming Shao, M.D, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Cancer Hospital/ Institute, Fudan University, Shanghai, Shanghai Municipality
  - Department of Breast Surgery, Cancer Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided